CLINICAL TRIAL: NCT01547832
Title: Metabolic Phenotyping of Subjects With Mutations Associated With Hereditary Parkinson's Disease
Brief Title: Mutations Associated With Parkinson s Disease
Status: Terminated | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120084; 12-H-0084
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08-27

CONDITIONS: Parkinson's Disease
Keywords: Cholesterol; Early Onset Parkinson's Disease; Fat Metabolism; Insulin Resistance; PARK2 Mutations
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Early-onset Parkinson's disease (EOPD) is more likely to be caused by gene mutations than Parkinson's disease that develops in older people. Studying these mutations may help find therapies for EOPD. Researchers want to study mutations on a gene called PARK2. These mutations prevent fat uptake into cells and may interfere with normal brain function. Researchers want to study fat and cholesterol in the body to look at the effects of these mutations on the body and brain.

Objectives:

- To study connections between genetic mutations and EOPD.

Eligibility:

* Individuals between 18 and 80 years of age with EOPD.
* Individuals between 18 and 80 years of age with no family history of Parkinson s disease.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will also be collected.
* Participants will have some or all of the following tests:
* Blood samples and tissue (skin and fat) biopsies
* Cell line development from these tissue samples to study the function of PARK2
* DEXA scan to measure body fat context using low dose x-rays
* Glucose and insulin tolerance testing to measure blood sugar levels.
* Treatment will not be provided as part of this protocol.

DETAILED DESCRIPTION:
The majority of subjects with the degenerative Parkinson s Disease present at around the age of 70 years. Other subjects develop this brain disease before the age of 40 years. This early onset presentation is more likely to have a direct genetic cause than the degenerative form of the disease. Our understanding of the genetic causes of early onset Parkinson s Disease may help us find therapies for both the genetic and more degenerative illnesses. Our laboratory has found that one of the genetic mutations associated with early onset Parkinson s Disease, in a gene called PARK2 results in impaired uptake of fat into cells. This may have detrimental effects in the brain, as the brain requires fat to make cholesterol and to send brain signals. A finding in mice lacking PARK2, is that they are resistant to diet induced diabetes and obesity and to fatty liver. These data suggests that the systemic and brain effects of low fat uptake may be opposing, with low fat uptake having a beneficial effect against risk factors such as obesity and diabetes but increasing the risk for brain diseases. To begin to test whether this is the case in subjects with PARK2 mutations we propose to test their fat uptake and glucose and insulin sensitivity.

ELIGIBILITY:
* INCLUSION CRITERIA:

Parkinson s Subjects:

Screening:

* Age 18 years to 80 years old with a history of early onset Parkinson disease (Presentation within the first five decades of life).
* Diagnosis of Parkinson disease or Parkinsonism
* Willingness and legal ability to give and sign informed study consent

Enrollment:

* Mutations in PARK2
* Willingness to travel to NIH for scheduled protocol studies

Control Subjects:

* Age 18 years to 80 years old with no history or family history of Parkinson disease.
* Willingness and legal ability to give and sign informed study consent
* Willingness to travel to NIH for scheduled protocol studies
* Willingness to have blood or tissue samples studied, and potentially stored for future research

EXCLUSION CRITERIA: <TAB>

Parkinson Subjects:

Screening:

* Subjects who are unable or unwilling to sign an informed consent subjects with genetic defects associated with other diseases including other neurologic syndromes.
* Subjects without medically treated diabetes who are unable/unwilling to undergo a glucose tolerance test

Enrollment:

- Pregnancy

Control Subjects

* Subjects who are unable or unwilling to sign an informed consent
* Subjects with genetic defects associated with other diseases including other neurologic syndromes.
* Pregnancy
* Medically treated diabetes
* Unable/unwilling to undergo a glucose tolerance test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02-27; Study Completion 2018-08-27

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Greenamyre JT, Hastings TG. Biomedicine. Parkinson's--divergent causes, convergent mechanisms. Science. 2004 May 21;304(5674):1120-2. doi: 10.1126/science.1098966. No abstract available. PMID 15155938
- [Background] Kitada T, Asakawa S, Hattori N, Matsumine H, Yamamura Y, Minoshima S, Yokochi M, Mizuno Y, Shimizu N. Mutations in the parkin gene cause autosomal recessive juvenile parkinsonism. Nature. 1998 Apr 9;392(6676):605-8. doi: 10.1038/33416. PMID 9560156
- [Background] Shimura H, Hattori N, Kubo Si, Mizuno Y, Asakawa S, Minoshima S, Shimizu N, Iwai K, Chiba T, Tanaka K, Suzuki T. Familial Parkinson disease gene product, parkin, is a ubiquitin-protein ligase. Nat Genet. 2000 Jul;25(3):302-5. doi: 10.1038/77060. PMID 10888878